CLINICAL TRIAL: NCT03348449
Title: A Retrospective Cohort Study of the Efficacy and Evolution of Comorbidities With the Combination of Raltegravir and Boosted Darunavir in Suppressed HIV-infected Patients With Intolerance or Toxicity to Nucleoside Analogues
Brief Title: Bitherapy With the Combination of Raltegravir and Darunavir (BIRDi)
Acronym: BIRDi
Status: Completed | Type: Observational
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jose L. Casado, Physician, Asociacion para el Estudio de las Enfermedades Infecciosas
Other Study IDs: EC 211/17
Record Dates: First submitted 2017-11-13; First posted 2017-11-20 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Comorbidities; HIV/AIDS
Keywords: HIV; Dual therapy; Comorbidities; Nucleoside analogues sparing-regimens
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Collection of data — Outcome of patients will be collected from charts to evaluate primary and secondary objectives

SUMMARY:
Retrospective cohort of virologically suppressed HIV-infected patients who received the combination of Raltegravir plus Darunavir boosted with cobicistat or ritonavir, as dual therapy, because or toxicity or intolerance to nucleoside analogues

DETAILED DESCRIPTION:
This is a retrospective cohort study including those HIV-infected patients who received the combination of raltegravir plus darunavir boosted with cobicistat or ritonavir as dual therapy, due to the existence of toxicity or intolerance to nucleoside analogues, to evaluate:

* efficacy, measured as percentage of patients free of virological failure after 48 and 96 weeks (ITT-e, snapchot analysis) and improvement in CD4+ count
* tolerance (rate of discontinuation and cause, and frequency of adverse events)
* evolution of different comorbidities (renal, bone, cardiovascular events)

Patients will included if they have received at least 1 dose of the dual therapy

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Older than 18 years
* To have received the combination of raltegravir plus boosted darunavir in patients with virological suppression (more than 6 months) after toxicity or intolerance to nucleoside analogues

Exclusion Criteria:

* Virological failure in the last 6 months previous to dual therapy
* Presence or suspicion of resistance to Darunavir (major mutations according to Meyer et al) or to Raltegravir (major mutations according to IAS list)
* Active hepatitis B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients with virological suppression but toxicity or intolerance to analogues who switched to the combination of Raltegravir plus boosted Darunavir
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who maintained virological suppression on treatment at 48 weeks after using this dual therapy | 48 weeks
  The number of patients who remained with virological suppression during the study at 48 weeks (ITT-exposed, snapchot analysis)

SECONDARY OUTCOMES:
Change in renal parameters at 48 weeks,for patients using dual therapy | 48 weeks
  Evaluation of renal parameters in patients changing to this dual therapy, considering the previous use of TDF or not.
Change in bone parameters (bone mineral density by Dual X-ray absorptiometry) during the study | 48 weeks
  Quantitative changes in bone mineral density (BMD) according to previous use of TDF and renal parameters
Change in cardiovascular risk (by using AHA score) for patients using dual therapy | 48 weeks
  Changes in lipid parameters will be assessed
Changes in inflammatory markers during the study, measured by the CD4/CD8 ratio | 48 weeks
  Those patients who received this dual therapy will be evaluated to determine changes in inflammatory biomarkers such as CD4/CD8 ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Ramon y Cajal Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No